CLINICAL TRIAL: NCT02617667
Title: A Phase 2, Multi-center, Randomized, Double-masked, Placebo (Vehicle)-Controlled Clinical Study With an Open Label Comparator Arm to Assess the Efficacy, Safety and Tolerability of Topical CyclASol® for Treatment of Dry Eye Disease
Brief Title: CyclASol for the Treatment of Moderate to Severe Dry-eye Disease (DED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novaliq GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CYS-002
Record Dates: First submitted 2015-11-25; First posted 2015-12-01 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-10

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporine; Excipients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- CyclASol Ophthalmic Solution 1 (Experimental): Cyclosporine A solution (dose-level 1) in vehicle
  Interventions: Drug: Cyclosporine A
- CyclASol Ophthalmic Solution 2 (Experimental): Cyclosporine A solution (dose-level 2) in vehicle
  Interventions: Drug: Cyclosporine A
- Placebo Ophthalmic Solution (Placebo Comparator): Vehicle only
  Interventions: Drug: Placebo
- Restasis (Active Comparator): Cyclosporine A 0.05% ophthalmic emulsion
  Interventions: Drug: Cyclosporine A

INTERVENTIONS:
Drug: Cyclosporine A — topical ocular, eye drops
  Other Names: Ciclosporin, CsA
  Arms: CyclASol Ophthalmic Solution 1; CyclASol Ophthalmic Solution 2; Restasis
Drug: Placebo — topical ocular, eye drops
  Other Names: Excipient
  Arms: Placebo Ophthalmic Solution

SUMMARY:
The objective of this study was to compare the safety, efficacy, and tolerability of two different dose levels of CyclASol Ophthalmic Solutions to placebo (vehicle) and Restasis for the treatment of the signs and symptoms of Dry Eye Disease (DED).

DETAILED DESCRIPTION:
This phase 2 study explored the safety, efficacy and tolerability of two CyclASol concentrations as one drop twice daily versus vehicle (placebo). In addition to the masked vehicle control arm, an open-label comparator arm consisting of Restasis was included.

The study explored a range of signs and symptoms of DED to gain an understanding of the possible treatment effects in comparison to vehicle and estimation of effect sizes. In line with current treatment guidelines, the proposed phase 2 population consisted of patients suffering from moderate to severe DED.

The primary treatment comparisons in this study were between the two CyclASol concentrations versus vehicle for the sign variable total corneal fluorescein staining and the symptom variable dryness severity visual analogue scale at day 113. All other comparisons between treatments groups were considered secondary analyses.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form and HIPAA (Health Insurance Portability and Accountability Act ) document
* Patient-reported history of dry eye in both eyes
* Current use of over-the-counter and/or prescription eye drops for dry eye symptoms
* Ability and willingness to follow instructions, including participation in all study assessments and visits

Exclusion Criteria:

* Women who are pregnant, nursing or planning a pregnancy
* Unwillingness to submit a blood pregnancy test at screening and at the last visit (or early termination visit) if of childbearing potential, or unwillingness to use acceptable means of birth control
* Clinically significant slit-lamp findings or abnormal lid anatomy at screening
* DED secondary to scarring or ocular or periocular malignancy
* History of herpetic keratitis
* Active ocular allergies or ocular allergies that are expected to be active during the study period
* Ongoing ocular or systemic infection at screening or baseline
* Wear of contact lenses within 3 months prior to screening or anticipated use of contact lenses during the study
* History of no response to previous topical Cyclosporine A and/or use of topical Cyclosporine A within 6 months prior to screening
* Intra-ocular surgery or ocular laser surgery within the previous 6 months, or have any planned ocular and/or lid surgeries over the study period
* Presence of an uncontrolled systemic disease
* Presence of a known allergy and/or sensitivity to the study drug or its components

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Kroesser, Dr.sc.hum., Study Director — Novaliq GmbH
Locations (4):
- United States (4):
  - CYS-002 Investigational Site, Newport Beach, California
  - CYS-002 Investigational Site, Lewiston, Maine
  - CYS-002 Investigational Site, Andover, Massachusetts
  - CYS-002 Investigational Site, Quincy, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wirta DL, Torkildsen GL, Moreira HR, Lonsdale JD, Ciolino JB, Jentsch G, Beckert M, Ousler GW, Steven P, Krosser S. A Clinical Phase II Study to Assess Efficacy, Safety, and Tolerability of Waterfree Cyclosporine Formulation for Treatment of Dry Eye Disease. Ophthalmology. 2019 Jun;126(6):792-800. doi: 10.1016/j.ophtha.2019.01.024. Epub 2019 Jan 28. PMID 30703441

RESULTS

PARTICIPANT FLOW:
Groups:
- CyclASol 0.05% Ophthalmic Solution: Blinded treatment arm. Cyclosporine A solution (0.05%) in vehicle. Topical ocular eye drops.
  1 drop in each eye, twice daily
- CyclASol 0.1% Ophthalmic Solution: Blinded treatment arm. Cyclosporine A solution (0.1%) in vehicle. Topical ocular eye drops.
  1 drop in each eye, twice daily.
- Placebo Ophthalmic Solution: Blinded treatment arm. Vehicle only. Topical ocular eye drops.
  1 drop in each eye, twice daily.
- Restasis: Active comparator, open label arm. Cyclosporine A 0.05% ophthalmic emulsion topical ocular eye drops.
  1 drop in each eye, twice daily.
Period: Overall Study
Arm/Group | CyclASol 0.05% Ophthalmic Solution | CyclASol 0.1% Ophthalmic Solution | Placebo Ophthalmic Solution | Restasis
Started | 51 | 51 | 52 | 53
Completed | 50 | 50 | 48 | 52
Not Completed | 1 | 1 | 4 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set included all randomized participants.
Groups:
- Restasis: Active comparator, open label arm . Cyclosporine A 0.05% ophthalmic emulsion topical ocular eye drops.
  1 drop in each eye, twice daily.
- Total: Total of all reporting groups
Arm/Group | CyclASol 0.05% Ophthalmic Solution | CyclASol 0.1% Ophthalmic Solution | Placebo Ophthalmic Solution | Restasis | Total
Number analyzed (Participants) | 51 | 51 | 52 | 53 | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (10.72) | 61.1 (12.29) | 61.3 (10.45) | 62.8 (11.20) | 62.4 (11.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 36 | 39 | 40 | 153
  Male | 13 | 15 | 13 | 13 | 54

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Visit 1) in Total Corneal Fluorescein Staining at 113 Days
Description: The primary analysis and objective of the study was to compare the two CyclASol groups versus vehicle (all blinded treatment arms) for one sign and one symptom endpoint. The open label active comparator arm was not included in the primary analysis to reduce the number of comparisons. The sign endpoint was the change from baseline in total corneal fluorescein staining at day 113. The cornea is divided into five regions: central, superior, inferior, nasal and temporal. Each region is graded from 0-3 based on the National Eye Institute scale, where 0 indicates no staining and 3 maximal staining. The total score is the sum of all these regions. The maximum score for each eye is 15.
Time Frame: Baseline to 113 Days
Population: Full analysis set population for worst eye. Worst eye: Eyes were eligible for analysis if they met all inclusion criteria. If both eyes qualified, the worst eye was taken as the eye with higher (worse) staining at Visit 1. If staining was the same, the right eye was selected as the worst eye.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CyclASol 0.05% Ophthalmic Solution | CyclASol 0.1% Ophthalmic Solution | Placebo Ophthalmic Solution
Number analyzed (Participants) | 51 | 51 | 52
units on a scale | -2.38 (2.156) | -2.10 (2.252) | -1.69 (2.619)

2. Primary Outcome: Change From Baseline (Visit 1) in Dryness Severity Visual Analog Scale (VAS) at 113 Days
Description: The primary analysis and objective of the study was to compare the the two CyclASol groups versus vehicle (all blinded treatment arms) for one sign and one symptom endpoint. The open label active comparator arm was not included in the primary analysis to reduce the number of comparisons. Furthermore, the open label character could have had an impact on patient reported outcomes. The symptom endpoint was the change from baseline in severity of dryness VAS at Day 113. Dryness severity was rated from 0 to 100%, where 0% corresponds to "no dryness" and 100% corresponds to "maximum dryness".
Time Frame: Baseline to 113 Days
Population: Full analysis set population for worst eye. Worst eye: Eyes were eligible for analysis if they met all inclusion criteria. If both eyes qualified, the worst eye was taken as the eye with higher (worse) staining at Visit 1. If staining was the same, the right eye was taken.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CyclASol 0.05% Ophthalmic Solution | CyclASol 0.1% Ophthalmic Solution | Placebo Ophthalmic Solution
Number analyzed (Participants) | 51 | 51 | 52
units on a scale | -11.00 (19.362) | -9.30 (27.832) | -13.85 (25.301)

ADVERSE EVENTS:
Time Frame: Adverse events reported were documented from the first dose of randomized study drug until the end of the last study day visit (day 113)
Groups:
- Placebo Ophthalmic Solution: Blinded treatment arm. Vehicle only Topical ocular eye drops.
  1 drop in each eye, twice daily.
Arm/Group | CyclASol 0.05% Ophthalmic Solution | CyclASol 0.1% Ophthalmic Solution | Placebo Ophthalmic Solution | Restasis
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51 | 0/52 | 0/53
Serious Adverse Events (participants affected / at risk) | 2/51 | 0/51 | 0/52 | 1/53
Other Adverse Events (participants affected / at risk) | 5/51 | 4/51 | 4/52 | 4/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CyclASol 0.05% Ophthalmic Solution (N=51) | CyclASol 0.1% Ophthalmic Solution (N=51) | Placebo Ophthalmic Solution (N=52) | Restasis (N=53)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CyclASol 0.05% Ophthalmic Solution (N=51) | CyclASol 0.1% Ophthalmic Solution (N=51) | Placebo Ophthalmic Solution (N=52) | Restasis (N=53)
Visual acuity reduced (Eye disorders) | 2 (2) | 4 (6) | 1 (2) | 4 (6)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days